CLINICAL TRIAL: NCT02571179
Title: Intranasal Fentanyl in Treatment of Labour Pain - Efficacy and Safety
Brief Title: Intranasal Fentanyl in Treatment of Labour Pain
Acronym: fentaobs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Admescope Ltd (Industry)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUH12_04_2010
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Labor Pain
Keywords: Labor pain; Fentanyl; Transmucosal
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Intranasal fentanyl
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intranasal fentanyl 50 microg/dose (Experimental): patient was given intranasal fentanyl 50 microg/dose up to 250 microg
  Interventions: Drug: intranasal fentanyl 50 microg dose up to 250 microg

INTERVENTIONS:
Drug: intranasal fentanyl 50 microg dose up to 250 microg — When contraction pain was ≥ 5/10 (numerical rating scale 0= no pain, 10= worst pain), the parturient was given a intranasal fentanyl 50 µg dose. After 15 minutes, if contraction pain was still ≥ 5/10, a second 50 µg intranasal dose was administered. Fentanyl was administered every 15 minute until contraction pain decreased to less than 5/10 or until the maximum fentanyl dose of 250 µg was administered.

SUMMARY:
Physiological changes during pregnancy are known to affect the pharmacokinetics of many drugs. Intranasal fentanyl is an interesting option for obstetric analgesia, but its use in pregnant patients has not been established. The investigators studied pharmacokinetics of intranasal fentanyl in labouring women and to subsequently evaluate the maternal and fetal safety after administration.

ELIGIBILITY:
Inclusion Criteria:

* healthy parturients with uncomplicated, single gestation pregnancies, full term (38-42 weeks of gestation) pregnancy, agreed to participate

Exclusion Criteria:

* a disease that might affect hepatic or renal function, contraindications to opioid analgesics, fetal growth retardation, signs of fetal asphyxia by cardiotocography, meconium stained amniotic fluid or placental insufficiency. The subjects should not have received fentanyl during the previous 14 days.

Not agreed to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Fentanyl maximum concentration | From the first intranasal fentanyl dose to birth of the newborn up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, PhD, Principal Investigator — Kuopio University Hospital, Kuopio, Finland
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: Undecided